CLINICAL TRIAL: NCT05308030
Title: Outcomes of Rivaroxaban and Aspirin in Patients With Lower Extremity Peripheral Arterial Disease After Endovascular Revascularization.
Brief Title: Outcomes of Rivaroxaban and Aspirin in PAD After Endovascular Revascularization
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Hassan Ahmed Elshimy, Doctor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Rivaroxaban in PAD after ER
Record Dates: First submitted 2022-03-24; First posted 2022-04-01 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Rivaroxaban; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Rivaroxaban and Aspirin — After the endovascular intervention, Anticoagulant therapy plus Antiplatelet therapy will be maintained (Aspirin 100 mg once daily and Rivaroxaban 2.5 mg twice daily) for 3 months, and then Aspirin alone indefinitely

SUMMARY:
Assessing the outcomes of using Rivaroxaban plus Aspirin in patients with Lower Extremity Peripheral Arterial Disease after Endovascular Revascularization

DETAILED DESCRIPTION:
Globally more than 200 million people suffer from peripheral artery disease (PAD), and the incidence is rising due to advancing age, high rates of smoking in certain regions of the world, and the rising incidence of type 2 diabetes.

PAD patients have wide-spread atherosclerosis and suffer a high risk of major cardiovascular (CV) events, with atherothrombosis as the underlying pathophysiologicmechanism. Symptomatic peripheral artery disease (PAD) is associated with a reduction in exercise capacity and quality of life and risk for tissue loss that is often treated with lower extremity revascularization (LER) to relieve symptoms and to prevent limb loss in a large portion of the population.

PAD is also associated with a heightened risk for major adverse cardiovascular and limb events.

LER is associated with a substantial increased risk of ischemic cardiovascular and limb events, including a 4-fold increased risk for acute limb ischemia (ALI), an ≈30% increased risk of myocardial infarction (MI), and an increased risk of rehospitalization after LER.

Observations from a large administrative database showed that patients with PAD after LER had an early heightened risk for ischemic limb events and a later increased risk for cardiovascular events.

Despite the common use of dual antiplatelet therapy after endovascular LER, this strategy is not supported by any Class 1A PAD guideline recommendations. Guidelines do give Class IIB recommendation for dual antiplatelet therapy for endovascular and surgical procedures (American and European) and Class IIA recommendation with Level of Evidence C for endovascular procedures (European),whereas use of dual antiplatelet therapy is discouraged by the American College of Chest Physicians Evidence-Based Clinical Practice Guidelines.

Recently Antiplatelet therapy with low-dose factor Xa inhibition with rivaroxaban 2.5 mg twice daily used in combination with aspirin have been shown to reduce ischemic cardiovascular and limb events in patients with stable PAD. In patients with PAD undergoing LER, the VOYAGER PAD trial (Vascular Outcomes Study of ASA Along With Rivaroxaban in Endovascular or Surgical Limb Revascularization for Peripheral Artery Disease) demonstrated superiority of the combination of rivaroxaban 2.5 mg twice daily plus aspirin 100 mg daily versus placebo plus aspirin on the composite outcome of ALI, major amputation of a vascular pathogenesis, cardiovascular death, ischemic stroke, or MI, but with a numeric increase in major TIMI (Thrombolysis in Myocardial Infarction) bleeding.

So, Investigators decided to assess the outcomes of using Rivaroxaban 2.5 mg twice daily plus Aspirin 100 mg in patients with lower extremity PAD after endovascular revascularization

ELIGIBILITY:
Inclusion Criteria:

* Age ≥40 .
* Documented moderate to severe symptomatic lower extremity atherosclerotic peripheral artery disease.
* Technically successful peripheral revascularization distal to the external iliac artery for symptomatic PAD (Peripheral artery disease) within the last 10 days prior to randomization.
* Subject is able and willing to comply with the protocol and to adhere to the follow-up requirements.
* Subject has provided written informed consent.

Exclusion Criteria:

* Subject's age less than 40.
* Patients undergoing revascularization for asymptomatic PAD or mild claudication without functional limitation of the index leg.
* Imminent or foreseeable amputation.
* Subject already had a major amputation on the affected extremity
* Subject has emergent ischemic lesion [such as gas forming infection].
* Subject has a known hypersensitivity or contraindication to anticoagulants, anti-platelets, or contrast media, which is not amenable to pre- treatment.
* Subject is not in the position to be primarily revascularized or refuses surgery.
* Acute embolic ischemia.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Patency | One year
  Determination of patency of the target limb is essentially by measuring Ankle brachial Index(ABI)